CLINICAL TRIAL: NCT05633251
Title: Using Reinforcement Schedules to Improve Carotenoid Levels, Reduce Fruit and Vegetable Waste, and Increase School Lunch Participation in El Paso
Brief Title: Using Reinforcement Schedules to Increase Fruit&Vegetable Intake, Reduce Waste, and Increase School Lunch Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico State University (Other)
Collaborators: Paso del Norte Health Foundation (Other); University of Texas (Other); Brigham Young University (Other); Ysleta Independent School District, El Paso (Unknown)
Responsible Party: Principal Investigator, Mihai Niculescu, Professor of Marketing, New Mexico State University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 12335 & 12324
Record Dates: First submitted 2020-12-27; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Behavioral Changes; Psychology, Social; Nutrition
Keywords: fruit, vegetable, food waste
MeSH Terms: interventions — Random Allocation

STUDY DESIGN:
Intervention Model Description: Number of participants below is best estimate of students exposed to the intervention based on school lunch participation rates.
Who Masked: Participant
Masking Description: Participants were not aware of the purpose of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School 1 (Experimental)
  Interventions: Behavioral: Variable (non-random) interval; Behavioral: Control
- School 2 (Experimental)
  Interventions: Behavioral: Variable (random) interval; Behavioral: Control
- School 3 (Experimental)
  Interventions: Behavioral: Variable (random) interval; Behavioral: Variable (random) interval with table tents

INTERVENTIONS:
Behavioral: Variable (random) interval — Using Variable (Random) Interval Reinforcement Schedules to Increase Fruit and Vegetable Intake, Reduce Fruit and Vegetable Waste, and Increase School Lunch Participation
  Arms: School 2; School 3
Behavioral: Variable (non-random) interval — Using Variable (Non-random) Interval Reinforcement Schedules to Increase Fruit and Vegetable Intake, Reduce Fruit and Vegetable Waste, and Increase School Lunch Participation
  Arms: School 1
Behavioral: Variable (random) interval with table tents — Using Variable (Random) Interval Reinforcement Schedules and Table Tents with Health-related Messages to Increase Fruit and Vegetable Intake, Reduce Fruit and Vegetable Waste, and Increase School Lunch Participation
  Arms: School 3
Behavioral: Control — No intervention
  Arms: School 1; School 2

SUMMARY:
Using small monetary rewards to reinforce healthy behaviors, such as the consumption of fruits and vegetables (F&V), the investigators tested fixed and variable reinforcement schedules in three middle schools.

The investigators measured carotenoid levels, as a biomarker of F&V intake, and F&V waste over the intervention time frame. The investigators also tracked the school lunch participation rates over time.

ELIGIBILITY:
Inclusion Criteria:

* students attending three participating middle schools (Ysleta Independent School District)

Exclusion Criteria:

* N/A

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1626 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2016-05-06 (Actual)

PRIMARY OUTCOMES:
Change in food waste | 24 weeks
  Daily fruit, vegetable, and other food waste (in lbs)
Change in fruit and vegetable intake | 12 weeks
  As measured by carotenoid level, a biomarker for total fruit and vegetable intake; measured before and after the intervention

SECONDARY OUTCOMES:
School lunch participation rates | 32 weeks
  Number of participants in the school lunch program

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Niculescu, PhD, Principal Investigator — New Mexico State University
Locations (1):
- Ysleta Independent School District, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No